CLINICAL TRIAL: NCT07063615
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the Safety and Efficacy of Scalp Cream for Symptom Relief and Microbiome Balance in Mild-moderate Seborrheic Dermatitis Patients.
Brief Title: A Clinical Study to Assess the Safety and Effectiveness of Scalp Cream for Symptom Relief and Microbiome Balance in Mild-moderate Seborrheic Dermatitis Patients.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Blossom Microbiotics LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NB250017-BM_1.0_30June
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Seborrheic Dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microbiome-Powered Cream (Experimental): Mode of Usage: Apply a generous amount of the cream to the affected area of the scalp. Gently part the hair using a wide-tooth comb or your fingertips to ensure direct contact with the scalp. Extend slightly beyond affected areas.
  Massage the cream gently into the skin until fully absorbed. Do not rinse off after application.
  Frequency: Apply twice daily - once after the morning shower and once before bedtime.
  Route of Administration: Topical Note For best results, the cream should be applied within 5 minutes of towel drying, while the scalp is slightly damp and soft. At night, ensure the cream is fully absorbed before lying down to avoid transfer to bedding materials like pillows or sheets.
  Interventions: Other: Microbiome-Powered Cream
- Placebo Hair Cream (Placebo Comparator): Mode of Usage: Apply a generous amount of the cream to the affected area of the scalp. Gently part the hair using a wide-tooth comb or your fingertips to ensure direct contact with the scalp. Extend slightly beyond affected areas.
  Massage the cream gently into the skin until fully absorbed. Do not rinse off after application.
  Frequency: Apply twice daily - once after the morning shower and once before bedtime.
  Route of Administration: Topical Note For best results, the cream should be applied within 5 minutes of towel drying, while the scalp is slightly damp and soft. At night, ensure the cream is fully absorbed before lying down to avoid transfer to bedding materials like pillows or sheets.
  Interventions: Other: Placebo Hair Cream

INTERVENTIONS:
Other: Microbiome-Powered Cream — Mode of Usage: Apply a generous amount of the cream to the affected area of the scalp. Gently part the hair using a wide-tooth comb or your fingertips to ensure direct contact with the scalp. Extend slightly beyond affected areas.
  Massage the cream gently into the skin until fully absorbed. Do not rinse off after application.
  Frequency: Apply twice daily - once after the morning shower and once before bedtime.
  Route of Administration: Topical Note Ensure the scalp is completely dry (within 5 minutes of towel-drying post-shower) before applying the cream. At night, ensure the cream is fully absorbed before lying down to avoid transfer to bedding materials like pillows or sheets.
  Arms: Microbiome-Powered Cream
Other: Placebo Hair Cream — Mode of Usage: : Apply a generous amount of the cream to the affected area of the scalp. Gently part the hair using a wide-tooth comb or your fingertips to ensure direct contact with the scalp. Extend slightly beyond affected areas.
  Massage the cream gently into the skin until fully absorbed. Do not rinse off after application.
  Frequency: Apply twice daily - once after the morning shower and once before bedtime.
  Route of Administration: Topical Note Ensure the scalp is completely dry (within 5 minutes of towel-drying post-shower) before applying the cream. At night, ensure the cream is fully absorbed before lying down to avoid transfer to bedding materials like pillows or sheets.
  Arms: Placebo Hair Cream

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the safety and efficacy of scalp cream for Symptom Relief and Microbiome Balance in mild-moderate Seborrheic Dermatitis patients.

DETAILED DESCRIPTION:
A total of 34 participants, including males and non-pregnant, non-lactating females aged between 20 and 55 years (inclusive) with a confirmed diagnosis of mild to moderate seborrheic dermatitis, will be enrolled in the study. Enrolment will be based on scalp skin type, which may be classified as dry, oily, or combination. Participants will be randomized in a 22:12 ratio to receive either Treatment A or Treatment B, respectively.

The study aims to complete evaluations for 30 participants-20 in the Treatment A group and 10 in the Treatment B group. The potential patient will be screened as per the inclusion and exclusion criteria only after obtaining the written informed consent from the patients. Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be called on the telephone by the recruiting department prior the enrolment visit. Patients will be told during screening (prior to enrolment) not to use any hair product including hair oil and hair cream on the study visit day.

There will be total of 4 visits during the study. The duration of the study will be 60 (+2 days) from the enrolment. Subjects will be instructed to visit the facility as per below visits.

Visit 01(Within 15 Days): Screening, ICD obtained. Visit 02 (Day 1): Enrolment, Baseline Evaluations, Treatment Usage, Post Treatment Usage Evaluations at 30 mins (T30 Mins).

Visit 03 (Day 30 +2 Days): Post-usage evaluation Visit 04 (Day 60 +2 Days): Post-usage evaluation and End of Study Telephonic Follow Up (Day 90 + 2 Days): A scripted telephonic follow-up schedule, will be implemented for Treatment group A to assess whether any seborrheic dermatitis (SD) symptoms have recurred following discontinuation of the treatment, 30 days after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-55 years (both inclusive) at the time of consent.
* Sex: Males and non-pregnant/non-lactating females (preferably equal number of males and females).
* Females of childbearing potential must have a self-reported negative urine pregnancy.
* Subject is in good general health as determined by the Investigator on the basis of medical history.
* Patients must have a confirmed diagnosis of mild to moderate scalp seborrheic dermatitis, with an ASFS score of at least 16 at the time of screening.
* The severity grade will be evaluated by the dermatologist using the ASFS scale during the clinical study.
* Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
* If the subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
* Patients are willing to give written informed consent and are willing to follow the study procedure.
* Patients who commit not to use any other medicated/ prescription shampoos/hair care products, any other hair growth products or hair colour or dye, other than the test treatment for the entire duration of the study.
* Patients who are having refrigerator at their home for storage of test treatment.
* Subject is willing and able to comply with study procedures, including all scheduled visits, treatment applications, and assessments.
* Subject is willing and able to follow the study directions, to participate in the study, returning for all specified visits.
* Subject must be able to understand and provide written informed consent to participate in the study.

Exclusion Criteria:

* Subject with known allergy or sensitization to test treatment ingredients.
* Subjects with a history of dermatological scalp conditions other than seborrheic dermatitis or dandruff (e.g., psoriasis, tinea capitis, lichen planopilaris).
* Subject who had taken topical treatment of dandruff for at least 4 weeks.
* Subject who had taken any systemic treatment for at least 3 months.
* Subject who have plans of shaving scalp hair during the study.
* Use of systemic or topical medications (e.g., corticosteroids, immunosuppressants, retinoids) known to affect skin or scalp within the past 3 months, or any medical history likely to interfere with study.
* Subject has any concurrent skin disease.
* History of alcohol or drug addiction.
* Subjects with an allergy to dairy products.
* Subjects with a history or current presentation of visibly inflamed, infected, or severely irritated scalp, or known sensitivity to topical or cosmetic products.
* Pregnant or breast feeding or planning to become pregnant during the study period.
* Use of antibiotics, antifungal medications, or oral/topical probiotics within the past 4 weeks
* History of chronic illness which may influence the cutaneous state.
* Subject have participated any clinical research study related to hair care products within past 3 months.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-02-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of the test treatments by assessing the change in Adherent Scalp Flaking Score (ASFS) from baseline, both within treatment group and between treatment groups. | To evaluate the effectiveness of the test treatments by assessing the change in Adherent Scalp Flaking Score (ASFS) from baseline on Day 01 and post usage of test treatment on Day 30 (+2 Days), Day 60 (+2 Days) and between treatment groups using ASFS s
  ASFS scale Mild: 16-24, Moderate :25-34, Severe : 35-80
To evaluate the effectiveness of the test treatment by assessing the change in flake coverage for quantification of adherent flakes from baseline, both within treatment group and between treatment groups. | from baseline on Day 01 and post usage of test treatment on Day 30 (+2 Days), Day 60 (+2 Days) and between treatment groups.
  change in flake coverage using CASLiteNova from 8 parts of the scal
To evaluate the effectiveness of the test treatment by assessing reduction in itching from baseline, both within treatment group and between treatment groups. | from baseline on Day 01 and post usage of test treatment at T30 mins on Day 01, Day 30 (+2 Days), Day 60 (+2 Days) and between treatment groups
  reduction in itching using VAS scale for itching
To evaluate the effectiveness of the test treatment by assessing change in Scalp Erythema Index from baseline, both within treatment group and between treatment groups. | from baseline on Day 01 and post usage of test treatment at T30 mins on Day 01, Day 30 (+2 Days), Day 60 (+2 Days) and between treatment groups.
  change in erythema Index using Mexameter® MX 18

SECONDARY OUTCOMES:
To evaluate the effectiveness of the test treatment by assessing change in scalp microbiome from baseline, both within treatment group and between treatment groups. | Samples will be collected at three time points: baseline on Day 01 (pre-treatment) and post usage of test treatment on Day 30 (+2 Days) and Day 60 (+2 Days) and between treatment groups.
  longitudinal changes in scalp microbiome composition and host response by collecting BD swabs and FLOQ swabs
To evaluate the effectiveness of the test treatment by assessing change in scalp barrier function from baseline, both within treatment group and between treatment groups. | baseline on Day 01 and post usage of test treatment at T30 mins on Day 01, Day 30 (+2 Days), Day 60 (+2 Days) and between treatment groups.
  change in scalp barrier function (Transepidermal Water loss) using Tewameter® TM Hex
To evaluate the effectiveness of the test treatment by assessing change in sebum production from baseline, both within treatment group and between treatment groups. | baseline on Day 01 and post usage of test treatment at T30 mins on Day 01, Day 30 (+2 Days), Day 60 (+2 Days) and between treatment groups.
  change in sebum production using Sebumeter® SM 815
To evaluate the effectiveness of the test treatment by assessing reduction in hair fall and non-adherent flake count from baseline, both within treatment group and between treatment groups. | baseline on Day 01 and post usage of test treatment on Day 30 (+2 Days), Day 60 (+2 Days) and between treatment groups.
  reduction in hair fall and non-adherent flake count using 60 second hair combing test
To evaluate the effectiveness of the test treatment by assessing change in general appearance of scalp from baseline, both within treatment group and between treatment groups. | baseline on Day 01 and post usage of test treatment at T30 mins on Day 01, Day 30 (+2 Days), Day 60 (+2 Days)
  change in general appearance of scalp skin i.e. Itchiness, redness, roughness, and scaliness
To evaluate the effectiveness of test treatment by assessing change in hair density and hair thickness from baseline, both within treatment group and between treatment groups. | on Day 01 and post usage of test treatment on Day 30 (+2 Days), Day 60 (+2 Days) and between treatment groups.
  assessing change in hair density and hair thickness using CASLiteNova
To evaluate the effectiveness of the test treatment by assessing treatment perception questionnaire through Quality of Life Questionnaire and PGIC questionnaire f | Day 01 and post usage of test treatment at T30 mins on Day 01, Day 30 (+2 Days), Day 60 (+2 Days) and between treatment groups.
  change in treatments perception questionnaire through Quality of Life Questionnaire using 5-point Likert scale and PGIC questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nayan Patel, Principal Investigator — NovoBliss Research Private Limited
Locations (1):
- NovoBliss Research Private Limited, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No